CLINICAL TRIAL: NCT03194061
Title: Hypofractionated Radiotherapy and Concurrent Cisplatin for Locally Advanced Head and Neck Cancer: A Feasibility Trial
Brief Title: Hypofractionated Radiotherapy and Concurrent Cisplatin for Head and Neck Cancer
Acronym: HIPOCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIPO CP.
Record Dates: First submitted 2017-04-24; First posted 2017-06-21 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2017-06

CONDITIONS: Radiotherapy; Complications
Keywords: chemotherapy; complication
MeSH Terms: interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypofractionated chemoradiation (Experimental): 20 fractions of 275cGy and concomitant weekly cisplatin 35mg/m2 x 4 cycles
  Interventions: Radiation: Hypofractionated Radiotherapy; Drug: Weekly cisplatin

INTERVENTIONS:
Radiation: Hypofractionated Radiotherapy — 20 fractions of 275cGy 5 days/week
Drug: Weekly cisplatin — Concomitant weekly cisplatin 35mg/m2 x 4 weeks

SUMMARY:
The aim of this study is to evaluate the feasibility of hypofractionated radiation therapy and concomitant chemotherapy with cisplatin for locally advanced head and neck cancer in a high volume brazilian center.

DETAILED DESCRIPTION:
To evaluate if concomitant cisplatin and hypofractionated radiation therapy wold be feasible in a brazilian population.

Patients eligibility criteria:

older than 18 years old Biopsy proven squamous cell carcinoma of oropharynx, larynx and hypopharynx. Stage III an IV, with no distant metastasis. ECOG performance status 0-2. Adequate renal and liver function. Good status for radical treatment

Treatment considered feasible if:

1. Patient receive at least 90% of radiation dose (18 of 20 fractions of 275cGy)
2. Patients receive at least 3 of 4 weekly cycles of cisplatin (35mg/m2)
3. Treatment length up to 35 days.
4. Grade 4 toxicity lower than 25%

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven squamous cell carcinoma of oropharynx, larynx and hypopharynx.
* Stage III an IV, with no distant metastasis.
* ECOG performance status 0-2.
* Adequate renal and liver function.
* Good status for radical treatment

Exclusion Criteria:

* Other oncologic treatment before
* Distant metastasis
* History of previous malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the rate of patient who could complete the treatment. | up to 5 years after patient accrual
  The treatment is considered completed when patients receive at least 90% of radiation dose (49,5Gy) with a cumulative cisplatin dose of 105mg/m2 or more (3 of 4 cycles) and the treatment duration is inferior to 35 consecutive days.
To evaluate the rate of participants with treatment-related adverse events | up to 5 years after patient accrual
  as assessed by investigators using the CTCAE v4.0 criteria

SECONDARY OUTCOMES:
Quality of life according to the EORTC C30 questionaire and EORTC H&N 35 (evaluated together) | up to 18 months from treatment
  Frequency and intensity of symptoms as described by patients before treatment (baseline), at the end of treatment, 1 month, 7 months and after 1 year following the treatment.
Response rate | up to 4 months after patient accrual
  as determined by investigators using RECIST v1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre A Jacinto, MD, Principal Investigator — Barretos Cancer Hospital; Andre Lopes Carvalho, Phd, Study Director — Barretos Cancer Hospital; Luciano Souza Viana, Phd, Study Chair — Barretos Cancer Hospital; Pedro de Marchi, Study Chair — Barretos Cancer Hospital; Eronides Salustiano Batalha, Study Chair — Barretos Cancer Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jacinto AA, Batalha Filho ES, Viana LS, De Marchi P, Capuzzo RC, Gama RR, Boldrini Junior D, Santos CR, Pinto GDJ, Dias JM, Canton HP, Carvalho R, Radicchi LA, Bentzen S, Zubizarreta E, Carvalho AL. Feasibility of concomitant cisplatin with hypofractionated radiotherapy for locally advanced head and neck squamous cell carcinoma. BMC Cancer. 2018 Oct 23;18(1):1026. doi: 10.1186/s12885-018-4893-5. PMID 30352576